CLINICAL TRIAL: NCT06464354
Title: Comparison of the Effect of Mammary Artery Harvesting Technique to Sternal Blood Supply Using Non-contact Dynamic Thermography
Brief Title: Comparison of the Mammary Harvesting Technique
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: KCHC-01-mammary artery; SGS25/LF/2023 (Other Grant/Funding Number: University of Ostrava)
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Heart Disease
Keywords: sternotomy; thermography; coronary bypass; LIMA; skeletonization technique
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LIMA - pedicle
  Interventions: Procedure: The mammary artery harvesting by the pedicle technique
- LIMA - skeletonised
  Interventions: Procedure: The mammary harvesting using the skeletonization technique
- Control group - LIMA not harvested
  Interventions: Procedure: No intervention

INTERVENTIONS:
Procedure: The mammary artery harvesting by the pedicle technique — The mammary artery harvesting by the pedicle technique was used in the LIMA pedicle study group.
  Groups: LIMA - pedicle
Procedure: The mammary harvesting using the skeletonization technique — The mammary harvesting using the skeletonization technique was used in the LIMA skeletonized study group.
  Groups: LIMA - skeletonised
Procedure: No intervention — No intervention was used in the control study group.
  Groups: Control group - LIMA not harvested

SUMMARY:
The skeletonization technique of left internal artery (LIMA) harvesting is reported as more spar-ing to the vascular supply of the sternum. Some studies report a greater length and greater flow of the graft additionally. The aim of our study was to measure the difference in post-op sternal blood supply compared to the pedicle harvesting technique and to measure the length and flow of the LIMA graft.

DETAILED DESCRIPTION:
A total of 90 patients were examined in a prospective randomized study. In 60 patients referred for coronary artery bypass grafting (CABG), LIMA was harvested, one-half (n=30) skeletonized, and one-half (n=30) with a pedicle. Thirty patients operated via sternotomy without LIMA harvesting (other procedures, for instance, valve surgery) were the control group. In patients undergoing LIMA harvest, harvest duration, graft length, and graft free flow were measured at defined arterial pressure. In all patients, the sternal blood flow was examined by active dynamic thermography (DIRT): first preoperatively and on 4th postoperative day. During this, the time of spontaneous rewarming of the skin surface after the application of a cold stimulus was measured in the caudal part of the sternum. The difference between postoperative and preoperative time was calculated and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery procedure via median sternotomy
* The left mammary artery (LIMA) harvesting for coronary bypass planned as a part of the operation - Group 1 and 2
* Other cardiac surgery procedures without the LIMA harvesting (valve surgery for instance) - Control group
* Signing of the informed consent

Exclusion Criteria:

* Emergent surgery
* Re-operation
* Re-sternotomy
* Thoracotomy approach
* Harvesting of both mammary arteries (BIMA)
* Endocarditis
* Ongoing non-cardiac infection
* Fever
* Circulatory failure
* Ongoing administration of catecholamines to patient
* Unsigned informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective cardiac surgery via sternotomy
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rewarming time difference | first preoperatively and on 4th postoperative day
  Duration of spontaneous rewarming of the skin surface of the caudal sternum after a cold stimulus, measured from 24°C to 27°C. Unit: seconds (s)

SECONDARY OUTCOMES:
Duration of the mammary graft harvesting | during surgery, immediately after the graft harvesting
  Time from the start of the harvesting to complete graft release. Unit: minute (min).
Length of the mammary artery graft | during surgery, immediately after the graft harvesting
  Length from the distance of the graft from the chest wall to its distal end. Unit: millimeter (mm).
Free outflow of the mammary artery | during surgery, just before the graft use
  After trimming the distal clip on the graft at an arterial pressure of 70 mmHg, free flow for 30 seconds, then multiplied by two. Unit: millilitre per minute (ml/min).

CONTACTS AND LOCATIONS:
Overall Officials: Radim Brát, Assoc.Prof.,MD,PhD,MBA, Study Chair — University Hospital Ostrava; Jiří Sieja, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravial-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Cheng K, Rehman SM, Taggart DP. A Review of Differing Techniques of Mammary Artery Harvesting on Sternal Perfusion: Time for a Randomized Study? Ann Thorac Surg. 2015 Nov;100(5):1942-53. doi: 10.1016/j.athoracsur.2015.06.087. Epub 2015 Sep 26. PMID 26410160
- [Background] Alom S, Yang N, Bin Saeid J, Zeinah M, Harky A. Harvesting internal mammary artery: a narrative review. J Cardiovasc Surg (Torino). 2020 Dec;61(6):790-801. doi: 10.23736/S0021-9509.20.11216-3. Epub 2020 Sep 4. PMID 32885924
- [Background] Lamy A, Browne A, Sheth T, Zheng Z, Dagenais F, Noiseux N, Chen X, Bakaeen FG, Brtko M, Stevens LM, Alboom M, Lee SF, Copland I, Salim Y, Eikelboom J; COMPASS Investigators. Skeletonized vs Pedicled Internal Mammary Artery Graft Harvesting in Coronary Artery Bypass Surgery: A Post Hoc Analysis From the COMPASS Trial. JAMA Cardiol. 2021 Sep 1;6(9):1042-1049. doi: 10.1001/jamacardio.2021.1686. PMID 34132753